CLINICAL TRIAL: NCT07246837
Title: A Randomized Controlled Trial of a Diagnostic Stewardship Intervention to Reduce Inappropriate Antibiotic Use for Urinary Tract Infections in Primary Care
Brief Title: Diagnostic Stewardship Intervention to Reduce Inappropriate Antibiotic Use for Urinary Tract Infections in Primary Care
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, LarisaGrigoryan, Associate Professor, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: H-53559; R01HS029489 (AHRQ)
Record Dates: First submitted 2025-11-19; First posted 2025-11-24 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Urinary Tract Infection(UTI); Antimicrobial Stewardship; Primary Care
Keywords: Urinary Tract Infection; UTI; Inappropriate Antibiotic Use; Diagnostic Stewardship; Antibiotic Resistance; Antimicrobial Stewardship; Primary Care; Randomized Controlled Trial
MeSH Terms: conditions — Urinary Tract Infections

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned in a 1:1 ratio to either the intervention group or the control group. The intervention group will receive a standardized educational tool, including a short video and flyer in English or Spanish, before urine collection to improve midstream clean-catch technique. The control group will receive usual care without additional education. All participants will collect urine samples using standard clinic materials, and samples will be processed according to routine laboratory protocols. The primary outcome is urine contamination status based on laboratory findings of epithelial cells or mixed flora. Secondary outcomes include antibiotic prescribing patterns, patient understanding of collection steps, and satisfaction with instructions. Randomization will be managed through REDCap. The study is open-label, and participation is voluntary with no impact on clinical care.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MSCC Educational Tool (Experimental): Participants receive a standardized educational tool prior to urine collection. This includes a short video and flyer in English or Spanish explaining proper midstream clean-catch technique. Materials are shown in the exam room before specimen collection.
  Interventions: Behavioral: MSCC Educational Tool
- Usual Care (No Intervention): Participants receive standard clinical care without additional educational materials. Urine collection follows routine clinic procedures.

INTERVENTIONS:
Behavioral: MSCC Educational Tool — A brief educational intervention (video + flyer) designed to improve urine collection technique and reduce contamination. Delivered in the patient's preferred language (English or Spanish) immediately before urine collection.
  Arms: MSCC Educational Tool

SUMMARY:
Urine culture is the most common microbiological test in the outpatient setting in the United States. Unfortunately, contamination during collection is prevalent and undermines test accuracy, leading to incorrect diagnosis, unnecessary treatment, wasted laboratory resources, and inflated costs. Unnecessary antibiotic treatment increases the risk of developing antimicrobial resistance, one of the most serious threats to patients and public health. The goal of this clinical trial is to test whether a bilingual (English and Spanish) educational intervention, an animated video and pictorial flyer, can reduce urine culture contamination and associated inappropriate antibiotic use in adult patients visiting safety-net primary care clinics.

The main questions it aims to answer are:

1. Does providing patients with a bilingual educational intervention reduce urine culture contamination rates?
2. Does the intervention lead to fewer unnecessary urinary antibiotic prescriptions?
3. Does providing patients with a bilingual educational intervention reduce contaminated urinalyses? Researchers will compare patients randomized to receive the educational intervention (video and flyer) to those receiving usual care to see if the intervention improves urine collection accuracy and reduces inappropriate antibiotic use. Participants will watch a short, animated video with step-by-step instructions for proper midstream clean-catch urine (MSCC) collection, receive a pictorial flyer (with stills from the video) reinforcing the instructions, and provide a urine sample for culture. Hypothesis: patients who receive the educational intervention will have: lower urine culture contamination rates (primary outcome), fewer urinary antibiotic prescriptions (secondary outcome), and fewer contaminated urinalyses (secondary outcome). The objectives are to (1) develop educational tools: Create an animated video and pictorial flyer with step-by-step urine collection instructions for women and men, developed through an iterative, stakeholder-engaged process, (2) assess acceptability: Use mixed methods (quantitative surveys and qualitative interviews) to evaluate and refine the tools for usability and cultural/linguistic appropriateness, and (3) test effectiveness: Conduct a randomized controlled trial to assess the intervention's impact on urine contamination rates, antibiotic prescribing, and patient satisfaction.

DETAILED DESCRIPTION:
Background: Urinary tract infections (UTIs) account for more than 10 million ambulatory visits annually in the United States and are the third-leading cause of outpatient antibiotic prescriptions. Gram-negative urinary pathogens collected from outpatients across all regions of the United States now exhibit antimicrobial resistance levels that exceed thresholds recommended for empiric treatment of UTIs. Accurate urine cultures are essential for guiding antibiotic therapy. Midstream clean-catch (MSCC) urine collection is the gold standard for obtaining urine specimens, yet contamination rates in outpatient settings range from 46% to 55% in the recent studies. Contamination leads to incorrect diagnoses, unnecessary antibiotic use, increased resistance, and higher healthcare costs. Prior interventions aimed at reducing contamination have had mixed results and lacked stakeholder engagement and effective educational modalities.

Significance: This study addresses Goal 3 of the National Action Plan for Combating Antibiotic-Resistant Bacteria and CDC priorities by improving diagnostic accuracy and reducing inappropriate antibiotic use. Our approach empowers frontline staff and targets a neglected area of outpatient diagnostic stewardship. Urine culture contamination is common, wasteful, and harmful, particularly for pregnant patients who are routinely screened for bacteriuria. Contamination obscures true infection or leads to overtreatment, increasing risks for antimicrobial resistance, adverse drug reactions, and healthcare costs. Our intervention will improve patient care and reduce waste of laboratory resources.

Innovation and Impact: The proposed research is innovative because it places nurses and medical assistants at the forefront of antimicrobial stewardship in primary care. The investigators will develop a bilingual, multicultural educational intervention that includes an animated instructional video and a pictorial flyer. These materials will provide step-by-step guidance for proper MSCC urine collection and will be designed with input from patients, nurses, and medical assistants to ensure cultural competence and clarity for individuals with low literacy. This approach represents a departure from previous interventions, which lacked stakeholder engagement and failed to reduce contamination rates effectively. By incorporating stakeholder feedback and using engaging visual formats, the investigators aim to create an intervention that is acceptable, appropriate, and feasible for diverse patient populations.

Specific Aims: Aim 1: Iteratively develop a bilingual, multicultural educational intervention to reduce urine contamination, with stakeholder and expert input. The intervention will include an animated instructional video and a flyer with pictorial instructions that will provide step-by-step guidance to patients for collecting an MSCC urine sample. Aim 2: Perform a pilot study to assess and improve the intervention's acceptability, appropriateness, and feasibility using mixed methods. The investigators will use a sequential explanatory design that includes a quantitative survey and qualitative interviews with stakeholders (patients, nurses, and medical assistants). Aim 3: Test the effectiveness of the intervention at reducing urine culture contamination via a randomized controlled trial. The investigators hypothesize that patients who are randomized to receive the intervention versus usual care will have lower culture contamination rates (primary outcome), fewer urinary antibiotic prescriptions (secondary outcome), and fewer contaminated urinalyses (secondary outcome). Investigators will also study intervention fidelity, usability, and patient satisfaction using mixed methods research.

Methodology: The study will be conducted in two safety-net and one private primary care clinics. The investigators will use a randomized controlled trial with parallel groups to compare the intervention to usual care. Eligible participants will be adults aged 18 years or older who are asked to provide a urine sample for culture or urinalysis. Patients with indwelling urinary catheters or those unable to view the video or read the flyer in English or Spanish will be excluded. Randomization will occur at the patient level using a secure electronic system managed through REDCap. Participants assigned to the intervention group will view the animated video and flyer in their preferred language before urine collection. Men will receive materials tailored for men, and women will receive materials tailored for women. Participants in the control group will receive usual care without additional education. The primary outcome is the proportion of contaminated urine cultures, defined as mixed flora, growth of non-uropathogens, or growth of three or more uropathogens. Secondary outcomes include antibiotic prescribing within seven days of urine culture results and contamination of urinalyses, defined as more than ten squamous epithelial cells per microscopic field. The investigators will also assess implementation results through exit interviews and surveys. The sample size for the trial is 252 patients (126 per arm). Data will be collected from electronic medical records, patient surveys, and qualitative interviews. All data will be securely stored and de-identified for analysis.

Next Steps/Implementation: If the intervention proves effective, future work will focus on disseminating the educational tools to other settings, such as emergency departments and long-term care facilities. This project will provide a scalable, resource-efficient approach to improving diagnostic accuracy, reducing unnecessary antibiotic use, and advancing antimicrobial stewardship in outpatient care.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥18 years) undergoing urine culture as part of routine outpatient care
* Able to provide informed consent
* English- and or Spanish-speaking.

Exclusion Criteria:

* Presence of a urinary catheter
* Inability to read and sign the informed consent
* Unable to follow study procedures (due to significant visual, auditory, physical or cognitive impairment).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 252 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2028-05-31 (Estimated)

PRIMARY OUTCOMES:
Urine Culture Contamination | Within 48 hours of specimen collection
  Presence of mixed flora, growth of non-uropathogens, or growth of three or more uropathogens in urine culture results.

SECONDARY OUTCOMES:
Contaminated Urinalysis Status | Within 24-48 hours of specimen collection
  Urine specimen will be considered contaminated if laboratory analysis reports 10 or more epithelial cells per high-power field.
Antibiotic Use | Within 7 days post-collection
  Antibiotic prescriptions associated with urine culture results.
Patient Understanding and Satisfaction | Immediately post-collection and after clinic visit.
  Exit interviews assessing comprehension of collection steps, intervention fidelity and usability, and satisfaction with instructions. This survey will be completed with patients who received the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Larissa Grigoryan, MD, PhD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared because participants did not provide consent for data sharing beyond the scope of this study, and sharing could compromise confidentiality despite de-identification efforts.

REFERENCES:
- [Background] Bekeris LG, Jones BA, Walsh MK, Wagar EA. Urine culture contamination: a College of American Pathologists Q-Probes study of 127 laboratories. Arch Pathol Lab Med. 2008 Jun;132(6):913-7. doi: 10.5858/2008-132-913-UCCACO. PMID 18517272
- [Background] Goebel MC, Trautner BW, Grigoryan L. The Five Ds of Outpatient Antibiotic Stewardship for Urinary Tract Infections. Clin Microbiol Rev. 2021 Dec 15;34(4):e0000320. doi: 10.1128/CMR.00003-20. Epub 2021 Aug 25. PMID 34431702
- [Background] Reekie D. Ending the misery of child dental decay. Br Dent J. 1999 Aug 28;187(4):174-6. doi: 10.1038/sj.bdj.4800234. PMID 10513105
- [Background] Gupta K, Grigoryan L, Trautner B. Urinary Tract Infection. Ann Intern Med. 2017 Oct 3;167(7):ITC49-ITC64. doi: 10.7326/AITC201710030. PMID 28973215